CLINICAL TRIAL: NCT01786343
Title: A Randomized Phase II Study of Two Schedules of Decitabine for Frontline Therapy of Older or Unfit Patients With Acute Myeloid Leukemia (AML)
Brief Title: Decitabine for Older or Unfit Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1017; NCI-2013-00463 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Leukemia
Keywords: Leukemia; Acute myeloid leukemia; AML; Response rates; Decitabine; Dacogen
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decitabine - 5 Day Regimen (Experimental): Decitabine 20 mg/m2 by vein daily for 5 days.
  Interventions: Drug: Decitabine
- Decitabine - 10 Day Regimen (Experimental): Decitabine 20 mg/m2 by vein daily for 10 days.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 20 mg/m2 by vein daily for either 5 or 10 days.
  Other Names: Dacogen

SUMMARY:
The goal of this clinical research study is to compare how well 2 different dosing schedules of decitabine may help control AML.

Decitabine is designed to damage the DNA (the genetic material) of cells, which may cause cancer cells to die.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 dose levels of decitabine based on when you join this study. If you are among the first 20 participants, you will have an equal chance of being in either group. If you enroll after that, you will have an increasingly higher chance (51-100%) of being assigned to the group that had better results, depending on how much better that treatment arm is.

Study Drug Administration:

Each cycle is about 4-8 weeks, depending on the doctor's decision. In this study you will receive induction therapy to try to control the disease and cause remission (this is when tests and/or the doctor cannot find signs of the disease).

If you are in Group 1, you will receive decitabine by vein over about 1 hour for 5 days.

If you are in Group 2, you will receive decitabine by vein over about 1 hour for 10 days.

If the disease is in remission, you may receive more cycles (called maintenance) to help keep the disease under control. If you are in Group 2, you will receive 5 day dosing during maintenance, or when the doctor thinks it is in your best interest.

Your dose schedule or dose level may be changed if the doctor feels it is in your best interest.

Study Visits:

The following tests and procedures will be performed:

* Blood (about 2-3 teaspoons) will be drawn 1-2 times weekly for first cycle, then every 2-4 weeks after that. After the 6th cycle or sooner if the doctor decides, this blood draw will be performed only 1 time per cycle.
* Every 1-3 cycles, you will have a bone marrow aspiration/biopsy to check the status of the disease. Blood (about 2-3 teaspoons) may also be drawn for genetic testing if the disease is in remission and the doctor thinks it is needed.

Length of Treatment:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation in this study will be over after the follow-up phone calls.

Follow-Up:

After you stop the study treatment, you will be called by phone twice a year and asked how you are feeling. The phone calls should last about 5 minutes each time.

This is an investigational study. Decitabine is FDA approved and commercially available for the treatment of myelodysplastic syndrome (MDS). Its use to treat AML is investigational.

Up to 100 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previously untreated AML (by the World Health Organization (WHO) criteria, i.e. >/= 20% blasts) Prior biologic therapies (such as growth factors) and targeted therapies administered for the treatment of prior myelodysplastic syndrome are allowed, with the exception of hypomethylating agents 5-azacytidine or decitabine. Patients must have been off such therapy for 1 week prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease. Hydroxyurea, and a single dose of cytarabine up to 3 g/m2, is permitted for control of counts prior to treatment.
2. Patients >/= 60 are eligible if not a candidate for standard cytarabine plus anthracycline chemotherapy as determined by Kantarjian's score (Appendix D) Patients younger than 60 may also be included if felt not to be a candidate for intensive anthracycline plus cytarabine based chemotherapy.
3. Performance 0-3 (ECOG).
4. Adequate liver function (Total bilirubin of < 2 mg/dl) unless due to hemolysis, leukemia organ infiltration or Gilbert's syndrome and renal function (creatinine < 2.5 mg/dl).
5. Signed informed consent

Exclusion Criteria:

1. Nursing and pregnant females. Female patients of childbearing potential and male patients should practice effective methods of contraception such as double barrier method. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Negative urine pregnancy test (women of childbearing potential)
2. Active and uncontrolled infections.
3. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, active significant other cancers requiring chemotherapy and/or radiation therapy within past 6 months (excluding non-melanoma skin cancer) or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-02-05 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Short NJ, Kantarjian HM, Loghavi S, Huang X, Qiao W, Borthakur G, Kadia TM, Daver N, Ohanian M, Dinardo CD, Estrov Z, Kanagal-Shamanna R, Maiti A, Benton CB, Bose P, Alvarado Y, Jabbour E, Kornblau SM, Pemmaraju N, Jain N, Gasior Y, Richie MA, Pierce S, Cortes J, Konopleva M, Garcia-Manero G, Ravandi F. Treatment with a 5-day versus a 10-day schedule of decitabine in older patients with newly diagnosed acute myeloid leukaemia: a randomised phase 2 trial. Lancet Haematol. 2019 Jan;6(1):e29-e37. doi: 10.1016/S2352-3026(18)30182-0. Epub 2018 Dec 10. PMID 30545576
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 2013 - April 2018
Pre-assignment Details: 74 participants were enrolled in the study, all participants completed the study.
Period: Overall Study
Arm/Group | Decitabine - 5 Day Regimen | Decitabine - 10 Day Regimen
Started | 28 | 46
Completed | 28 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine - 5 Day Regimen | Decitabine - 10 Day Regimen | Total
Number analyzed (Participants) | 28 | 46 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 25 | 46 | 71
Age, Continuous [Median (Full Range); unit: years] | 77 [57 to 85] | 78 [65 to 94] | 78 [57 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 16 | 32 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 22 | 36 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 28 | 46 | 74

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Response is defined as Complete Response (CR) + Partial Remission (PR) + Complete Remission with incomplete recovery (CRi) + Clinical Benefit. CR is the normalization of the peripheral blood and bone marrow with </= 5% bone marrow blasts, a peripheral blood granulocyte count >/= (1.0 x 10^9/L, and a platelet count >/= 100 x 10^9/L). PR is the same as CR except for the presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment. CRi meets all criteria for CR except for platelet recovery to >100 x 10^9/L and/or granulocyte count > (1.0 x 10^9/L). Clinical benefit is platelets increase by 50% and to above 30 x 10^9/L untransfused (if lower than that pretherapy); or granulocytes increase by 100% and to above 10^9/L (if lower than that pre-therapy); or hemoglobin increase by 2 g/dl; or transfusion independent; or splenomegaly reduction by > 50%; or monocytosis reduction by > 50% if pretreatment > 5 x 109/L.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine - 5 Day Regimen | Decitabine - 10 Day Regimen
Number analyzed (Participants) | 28 | 46
Participants | 12 | 19

2. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Decitabine - 5 Day Regimen | Decitabine - 10 Day Regimen
Number analyzed (Participants) | 28 | 46
Months | 5.5 [2.1 to 11.7] | 6.0 [1.9 to 11.7]

3. Secondary Outcome: Response Duration
Description: The date of response to date of loss of response or last follow-up. Response is defined as Complete Response (CR) + Partial Remission (PR) + Complete Remission with incomplete recovery (CRi) + Clinical Benefit. CR is the normalization of the peripheral blood and bone marrow with </= 5% bone marrow blasts, a peripheral blood granulocyte count >/= (1.0 x 10^9/L, and a platelet count >/= 100 x 10^9/L). PR is the same as CR except for the presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment. CRi meets all criteria for CR except for platelet recovery to >100 x 10^9/L and/or granulocyte count > (1.0 x 10^9/L). Clinical benefit is platelets increase by 50% and to above 30 x 10^9/L untransfused (if lower than that pretherapy); or granulocytes increase by 100% and to above 10^9/L (if lower than that pre-therapy); or hemoglobin increase by 2 g/dl; or transfusion independent; or splenomegaly reduction by > 50%; or monocytosis reduction by > 50% if pretreatment
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Decitabine - 5 Day Regimen | Decitabine - 10 Day Regimen
Number analyzed (Participants) | 28 | 46
Months | 9.4 [5.6 to 17.9] | 6.4 [2.8 to 12.4]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Decitabine - 5 Day Regimen | Decitabine - 10 Day Regimen
All-Cause Mortality (participants affected / at risk) | 5/28 | 16/46
Serious Adverse Events (participants affected / at risk) | 20/28 | 37/46
Other Adverse Events (participants affected / at risk) | 22/28 | 39/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine - 5 Day Regimen (N=28) | Decitabine - 10 Day Regimen (N=46)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (2)
Bactreamia (Infections and infestations) | 2 (2) | 0 (0)
Blood Clot (Vascular disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 3 (4)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
CVA Left Hemiparesis (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 16 (16)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Edema (General disorders) | 0 (0) | 3 (3)
Elevated Troponins (Investigations) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0)
Generalized Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hemorrhage CNS (Nervous system disorders) | 1 (1) | 0 (0)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Left Neck Mass - Lymph nodes (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 3 (3) | 7 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenic Fever (Infections and infestations) | 8 (10) | 13 (21)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Pseudomonas (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine - 5 Day Regimen (N=28) | Decitabine - 10 Day Regimen (N=46)
Hyperbilirubinemia (Investigations) | 2 (2) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 3 (3)
Elevated Creatinine (Investigations) | 5 (6) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Edema limb (General disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 6 (7) | 6 (12)
Neutropenic Fever (Infections and infestations) | 8 (9) | 14 (20)
Hypotension (Cardiac disorders) | 1 (1) | 3 (3)
Infection (Infections and infestations) | 2 (3) | 7 (8)
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (8)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (4)
Opportunistic Infection (Infections and infestations) | 7 (8) | 13 (13)
Pain (General disorders) | 2 (2) | 10 (11)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT01786343/Prot_SAP_000.pdf